CLINICAL TRIAL: NCT04720885
Title: Management of Large Retained Products of Conception (> 4 cm): Need for an Standardized Procedure.
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07879-ADP
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Placenta, Retained; Placenta; Retention, Fragments, Complicating Puerperium, Without Hemorrhage; Placenta; Retention, Fragments, Complicating Puerperium (Delayed Hemorrhage); Pregnancy Related; Hysteroscopy / Methods; Retrospective Studies; Vacuum Curettage
MeSH Terms: conditions — Placenta, Retained

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a placental remnant in medical history
  Interventions: Procedure: kind of surgery

INTERVENTIONS:
Procedure: kind of surgery — hysteroscopy, curettage, other

SUMMARY:
Collection of relevant data form patients who were treated in the Ghent University Hospital in the context of a placental remnant lager than 4 cm, performing statistical analyzes on the collected data, reviewing the literature on the subject and formulation of a recommendation for treatment of these large placental remnants.

ELIGIBILITY:
Inclusion Criteria:

* retained products of conception larger than 4 cm in largest dimension

Exclusion Criteria:

* retained products of conception 4 cm or smaller in largest dimension

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with a placental remnant in medical history.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Hysteroscopy | time of surgery
  Kind of surgery to remove retained products of conception
Vacuum Curettage | time of curettage
  Kind of surgery to remove retained products of conception
Polyp forceps | time of surgery
  Surgical instrument to remove retained products of conception
Prostaglandines | time of surgery
  Pharmacological agent to remove retained products of conception

CONTACTS AND LOCATIONS:
Overall Officials: Tjalina Hamerlynck, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium